CLINICAL TRIAL: NCT05250102
Title: Accuracy and Precision of Peripheral Capillary Oxygen Saturation of Reprocessed Pulse Oximetry Sensors Compared to Oxygen Saturation in Arterial Blood Samples Assessed by CO-oximetry in Neonates
Brief Title: Neonatal Pulse Oximetry Sensor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MED-2020-DIV65-001
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pulse oximeter sensor readings (Other): Subjects who satisfy all of the inclusion criteria will be eligible to participate in the study, will receive intervention (the Masimo and Nellcor sensors, and their arterial blood sample will be taken in the normal course of care). This is a single arm study. Those who don't meet the inclusion/ exclusion criteria won't be eligible to participate.
  Interventions: Device: Pulse oximeter sensors

INTERVENTIONS:
Device: Pulse oximeter sensors — Pulse oximeter reading will be compared to CO-oximeter reading.

SUMMARY:
To validate the SpO2 accuracy, bias, and precision of Medline's reprocessed pulse oximetry sensors as compared to SaO2 in arterial blood samples as assessed by CO-oximetry in neonates.

DETAILED DESCRIPTION:
Pulse oximetry helps in measuring peripheral capillary oxygen saturation (SpO2) continuously and non-invasively, and provides an indirect measurement of arterial oxygenation (SaO2) based on the red and infrared light-absorption characteristics of oxygenated and deoxygenated hemoglobin. Uses of pulse oximetry include detection of hypoxia, avoidance of hyperoxia, titration of fractional inspired oxygen, and enabling weaning from mechanical ventilation. Arterial blood gas (ABG) analysis, such as by the use of CO-oximeter, provides a direct measurement of SaO2. However, ABG analysis requires time, expense, and arterial access. Therefore, this study aims to validate the SpO2 accuracy of pulse oximetry sensors (manufactured by Nellcor and Masimo, and reprocessed by Medline Industries, LP) in neonates as compared to ABG measurements as part of their clinical standard of care (SOC), as assessed by CO-oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are postnatal 28 days or younger (neonates)
* Subjects who are likely to receive one or more ABG measurements as part of their clinical SOC
* Subjects who weigh less than 5 Kg (weight range for thesensors)

Exclusion Criteria:

* Subjects with current signs and symptoms of a clinically significant Patent Ductus Arteriosus (PDA) combined with a current or planned arterial line placement which will affect the validity of the co-oximetry measurement
* Subjects with physical malformation of hands, fingers, feet, or toes that would limit the ability to place sensors for this study
* Subjects judged by the Principal Investigator (PI) to be inappropriate for participation in this study
* Subjects for whom placing a pulse oximeter will cause dermatological issues (e.g. allergic to foam rubber or adhesive tape)

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Eastern Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ascha M, Bhattacharyya A, Ramos JA, Tonelli AR. Pulse Oximetry and Arterial Oxygen Saturation during Cardiopulmonary Exercise Testing. Med Sci Sports Exerc. 2018 Oct;50(10):1992-1997. doi: 10.1249/MSS.0000000000001658. PMID 29771822
- [Background] Dawson JA, Davis PG, O'Donnell CP, Kamlin CO, Morley CJ. Pulse oximetry for monitoring infants in the delivery room: a review. Arch Dis Child Fetal Neonatal Ed. 2007 Jan;92(1):F4-7. doi: 10.1136/adc.2006.102749. No abstract available. PMID 17185428
- [Background] Bland JM, Altman DG. Agreement between methods of measurement with multiple observations per individual. J Biopharm Stat. 2007;17(4):571-82. doi: 10.1080/10543400701329422. PMID 17613642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: a total of 23 neonates were recruited for the study, with 1-3 measurement pairs taken for each subject and each pulse oximetry sensor, for a total of 2, 4, or 6 measurement pairs per subject.
Period: Overall Study
Arm/Group | Pulse Oximeter Sensor Readings
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 23 to 29 weeks
Arm/Group | Pulse Oximeter Sensor Readings
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 23.6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 14
  White - Non Hispanic or Latino | 8
  Hispanic or Latino | 1

OUTCOME MEASURES:

1. Primary Outcome: Bland-Altman Analysis for Nellcor Pulse Oximeter
Description: BIAS Measurement and 95% confidence interval calculated using a Bland-Altman plot (mean vs. difference of SaO2 and SpO2) and an error plot (SaO2 vs. difference of SaO2 and SpO2) were generated. The B&A plot analysis is a simple way to evaluate a bias between the mean differences, and to estimate an agreement interval, within which 95% of the differences of the second method, compared to the first one, fall. Data can be analyzed both as unit differences plot and as percentage differences plot. We ran a percentage mean difference plot.
Time Frame: 15 episodic minutes
Population: all neonates participating in the study
Measure: Mean (95% Confidence Interval); unit: percentage of difference in mean
Groups:
- Sensor Massimo or Nellcor: Each participant wore massimo and nellcor sensors at the same time. Readings were taken from each sensor.
Arm/Group | Sensor Massimo or Nellcor
Number analyzed (Participants) | 23
percentage of difference in mean
  Bias Massimo | .151 [-.361 to .662]
  Bias Nellcor | .434 [-.149 to 1.017]

ADVERSE EVENTS:
Time Frame: Neonates enrolled in the study were monitored until discharge from the hospital, on average for 2 weeks.
Arm/Group | Pulse Oximeter Sensor Readings
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT05250102/Prot_SAP_000.pdf